CLINICAL TRIAL: NCT06476132
Title: Belumosudil to Block Chronic Lung Allograft Dysfunction (CLAD) in High Risk Lung Transplant Recipients: A Randomized, Multicenter, Double Blind, Placebo-Controlled Trial (CTOT-47)
Brief Title: Belumosudil to Block Chronic Lung Allograft Dysfunction (CLAD) in High Risk Lung Transplant Recipients
Acronym: CLAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT CTOT-47
Record Dates: First submitted 2024-05-08; First posted 2024-06-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Lung Transplant
Keywords: Lung Transplant; Belumosudil; CLAD; Acute Rejection; Lymphocytic Bronchiolitis; Organizing Pneumonia; Acute Lung Injury
MeSH Terms: conditions — Organizing Pneumonia; Acute Lung Injury | interventions — belumosudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belumosudil plus maintenance IS (Experimental): Eligible lung transplant recipients who experience a qualifying biopsy 60 to 550 days posttransplant will be randomized into the study. 200 mg of Belumosudil (increased to 200 mg twice daily in participants receiving concurrent strong CYP3A inducers or PPIs) + maintenance IS will be administered daily for one year from randomization.
  Interventions: Drug: Belumosudil
- Placebo + maintenance IS (Placebo Comparator): Eligible lung transplant recipients who experience a qualifying biopsy 60 to 550 days posttransplant will be randomized into the study. Placebo plus maintenance immunosuppression (IS) will be administered for one year
  Interventions: Drug: Placebo for Belumosudil

INTERVENTIONS:
Drug: Belumosudil — Participants will receive Belumosudil 200 mg daily (increased to 200 mg twice daily in participants receiving concurrent strong CYP3A inducers or PPIs) + maintenance IS for a duration of one year from randomization.
  Arms: Belumosudil plus maintenance IS
Drug: Placebo for Belumosudil — Participants will receive Placebo for Belumosudil 200 mg daily (increased to 200 mg twice daily in participants receiving concurrent strong CYP3A inducers or PPIs) + maintenance IS for a duration of one year from randomization.
  Arms: Placebo + maintenance IS

SUMMARY:
The purpose of this study is to see if taking the study drug, Belumosudil, for 52 weeks in addition to your usual care and medication, will prevent Chronic Lung Allograft Dysfunction (CLAD) in participants who have a lung biopsy that shows evidence of rejection or inflammation to the transplanted lung(s). For this study, biopsies that show evidence of Acute Rejection (AR), Lymphocytic Bronchiolitis (LB), Organizing Pneumonia (OP) or Acute Lung Injury (ALI) are referred to as "Qualifying Biopsies"; patients who had evidence of one or more of these conditions on a recent biopsy are eligible for enrollment in this study. Belumosudil is an investigational drug that blocks a molecule in the body that reduces inflammation and scarring and may play a role in the development and progression of CLAD. Belumosudil is a drug approved by the FDA to treat adults and children 12 years and older with chronic graft-versus-host disease (cGVHD), a condition with some similarities to CLAD.

The primary objective it to determine the efficacy of treatment with Belumosudil + maintenance immunosuppression (IS) versus placebo + maintenance IS on preventing the subsequent development of probable or definite CLAD, lung retransplant, or death.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent or guardian must be able to understand the purpose of the study, willing to participate, sign the informed consent, and if applicable assent.
2. Single or bilateral lung transplant recipient age ≥ 12 years
3. A qualifying biopsy obtained 60 to 550 days after lung transplant with evidence of allograft injury histology; a qualifying biopsy must have one or more of the following features alone or in combination: Acute Rejection (AR), Lymphocytic Bronchiolitis (LB), Organizing Pneumonia (OP), or Acute Lung Injury (ALI). The presence of any grade AR (A1 or greater) or LB (B1 or greater) qualifies for inclusion
4. Females of reproductive potential and males with female partners of reproductive potential must agree to use effective contraception during treatment with belumosudil or placebo and for at least 3 months after the last dose. Participants must agree to refrain from donating or cryopreserving sperm, eggs (ova or ovocytes) for the purpose of reproduction during treatment with belumosudil or placebo and for at least 3 months after the last dose.
5. Meeting hematologic laboratory criteria: absolute neutrophil count (ANC) >= 0.5 x 10(9)/L and platelet count >= 50 x 10(9)/L within 30 days of enrollment
6. Meeting all blood chemistry laboratory criteria: aspartate aminotransferase (AST) or alanine transaminase (ALT) < 2x upper limit of normal (ULN), bilirubin < 1.5x ULN unless due to Gilbert's syndrome, estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m2 within 30 days of enrollment
7. Cytomegalovirus (CMV) polymerase chain reaction (PCR) negative within 30 days of enrollment
8. In the absence of contraindications, must have received adult vaccinations or documented immunity as outlined in current National Institute of Allergy and Infectious Diseases (NIAID) Division of Allergy, Immunology, and Transplantation (DAIT) Guidance for Patients in Transplant Trials
9. Receiving Calcineurin Inhibitor (CNI)-based maintenance Immunosuppression (IS) regimen

Exclusion Criteria:

1. Multi-organ transplants involving more than one organ type (e.g., heart-lung)
2. Prior organ transplant or prior bone marrow transplant/hematopoietic stem cell transplantation
3. Greater than 120 days after a qualifying biopsy
4. Clinical AMR prior to enrollment. Subclinical AMR is permitted if 90 days or greater prior to enrollment.
5. Diagnosed with probable or definite CLAD according to International Society for Heart and Lung Transplantation (ISHLT) guidelines prior to enrollment.
6. Posttransplant treatment with anti-thymocyte globulin within 30 days or alemtuzumab or any other prohibited medication within 90 days prior to enrollment.
7. Epstein-Barr virus (EBV) seronegative recipient who received EBV positive donor lung(s).
8. Treatment with any other investigational pharmacologic agent within 30 days prior to enrollment.
9. Significant active uncontrolled infection which, in the opinion of the investigator, would place the participant at increased risk.
10. Current use of sirolimus or everolimus.
11. Recipient human immunodeficiency virus (HIV) positive.
12. Recipient Hepatitis B surface antigen positive or Hepatitis B core antibody positive.
13. Received lung(s) from a donor with known Hepatitis B virus (HBV) including Hepatitis B core antibody positive donors.
14. Recipient history of Hepatitis C, Hepatitis C seropositive, or received lung(s) from a donor with known Hepatitis C (participants who have 3 months of documented consecutive undetected Hepatitis C virus PCR after treatment or spontaneous clearance will not be excluded).
15. History of clinically significant surgical factors (such as phrenic nerve damage, transplant lung resection, chest wall surgery), or mechanical factors (such as posttransplant airways disease including bronchial dehiscence, stenosis, dilation, or stent placement, pleural disease) that impedes lung function.
16. Past or current medical problems, psychosocial concerns, or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose undue risk from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.
17. Pregnant or breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to the first occurrence of probable or definite CLAD (per ISHLT 2019 standard defined criteria), lung retransplant, or death | From randomization until study completion - scheduled assessments: minimum of 1 year, maximum of 3 years
  Probable CLAD is defined as a >= 20% decline in Forced Expiratory Volume in 1 Second (FEV1) compared to the baseline value on 2 measurements taken at least 3 weeks apart and after exclusion or adequate treatment of potential secondary causes of allograft dysfunction.
  The baseline FEV1 value is defined as the average of the 2 best posttransplant FEV1s taken at least 3 weeks apart

SECONDARY OUTCOMES:
Time from randomization to first occurrence of probable or definite CLAD (per ISHLT 2019 standard defined criteria) or lung retransplant | From randomization until study completion - scheduled assessments: minimum of 1 year, maximum of 3 years
  Definite CLAD is a sustained decline in pulmonary function as defined by a persistent decline in lung function meeting the definition of probable CLAD but sustained for a duration of at least 3 months
Time from randomization to death | From date of randomization until the date of death, through study completion; participants are scheduled to be assessed for a minimum of 1 year up to a maximum of 3 years
Time from randomization to first occurrence of the specific CLAD phenotypes of Restrictive Allograft Syndrome (RAS), Bronchiolitis Obliterans Syndrome (BOS), mixed, or undefined | From date of randomization until study completion - scheduled assessments: minimum of 1 year, maximum of 3 years
Frequency of Acute Rejection (AR) | Number of AR events occurring from date of randomization until date of end of treatment visit, an average of 1 year
Frequency of Lymphocytic Bronchiolitis (LB) | Number of LB events occurring from date of randomization until date of end of treatment visit, an average of 1 year.
Frequency of Organizing Pneumonia (OP) | Number of OP events occurring from date of randomization until date of end of treatment visit, an average of 1 year.
Frequency of Acute Lung Injury (ALI) | Number of ALI events occurring from date of randomization until date of end of treatment visit, an average of 1 year.
Rate of change in lung function measures (forced expiratory volume [FEV1] and forced vital capacity [FVC]) | Rate of change occurring from date of randomization until date of end of treatment visit, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M. Palmer, M.D., M.H.S., Study Chair — Duke University Medical Center: Transplantation
Locations (10):
- United States (10):
  - University of California, Los Angeles (Site #: 71123), Los Angeles, California
  - Johns Hopkins (Site #: 71119), Baltimore, Maryland
  - University of Minnesota (Site 71151), Minneapolis, Minnesota
  - Washington University (Site #: 71157), St Louis, Missouri
  - NYU Langone Health (Site #: 71177), New York, New York
  - Duke University (Site #: 71139), Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center (Site #: 71017), Cincinnati, Ohio
  - Cleveland Clinic (Site #: 71101), Cleveland, Ohio
  - University of Pennsylvania (Site #: 71111), Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center (Site #: 71174), Nashville, Tennessee

REFERENCES:
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/